CLINICAL TRIAL: NCT07318324
Title: Phase Ib Study of Avutometinib, Defactinib, and Everolimus in RAS Pathway Mutant Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1174; NCI-2025-09476 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-12-29; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Phase IB; Avutometinib; RAS Pathway; Endometrial
MeSH Terms: interventions — defactinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): To be administered per dose level during Days 1-21
  Interventions: Drug: Avutometinib; Drug: defactinib; Drug: Everolimus
- Dose Expansion (Experimental): To be administered per identified RP2D during Days 1-2
  Interventions: Drug: Avutometinib; Drug: defactinib; Drug: Everolimus

INTERVENTIONS:
Drug: Avutometinib — Given by PO
Drug: defactinib — Given by PO
Drug: Everolimus — Given by PO

SUMMARY:
To find the recommended dose of the combination of avutometinib, defactinib, and everolimus in patients with endometrial cancer that is recurrent and has abnormal RAS activity. The safety and effects of this combination will also be studied.

DETAILED DESCRIPTION:
Primary Objectives To identify the recommended phase 2 dosing (RP2D) of the combination of avutometinib, defactinib and everolimus in participants with recurrent, RAS pathway mutant endometrial cancer.

Secondary Objectives To evaluate the tolerability of the RP2D of avutometinib, defactinib and everolimus including dose limiting toxicities that occur during cycle 1.

ELIGIBILITY:
Eligibility Criteria

1. Participants must have histologically or cytologically confirmed recurrent RAS mutant endometrial cancer. RAS pathway gene activating mutations include KRAS, NRAS, HRAS, BRAF, MEK1, and MEK2 activating mutations. Any endometrial histology is permitted, including endometrioid, clear cell, mesonephric, and serous.
2. Participants must have received prior immune checkpoint inhibition treatment alone or in combination.
3. Unlimited prior systemic therapies are allowed, including any number of prior MEK inhibitor therapies is allowed.
4. Ability to understand and the willingness to sign a written informed consent document.
5. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
6. ECOG performance status of 0-1
7. The effects of avutometinib and defactinib on the developing human fetus are unknown. For this reason, women of child-bearing potential must have a negative urine or serum pregnancy test within 72 hours of starting study and agree to use adequate contraception prior to study entry, for the duration of study participation, and for 3 months after the last does of study drug. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

   * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
   * History of hysterectomy or bilateral salpingo-oophorectomy.
   * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
   * History of bilateral tubal ligation or another surgical sterilization procedure.

   The use of hormonal contraception methods is not recommended for this study. Approved methods of birth control are as follows: Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
8. Participants must have measurable disease as defined by RECIST v1.1
9. Age ≥18 years.
10. Participants must have adequate organ and marrow function as defined below:

    absolute neutrophil count ≥1,000/mcL platelets ≥100,000/mcL total bilirubin ≤ 1.5x institutional ULN AST(SGOT)/ALT(SGPT) ≤3× institutional ULN creatinine clearance > 50 ml/min hemoglobin > 9 g/dL If a red blood cell transfusion or erythropoiesis-stimulating agent has been administered the hemoglobin must remain stable and ≥ 9 g/dL for at least 1 week prior to first dose of study intervention.
11. Creatine phosphokinase (CPK) ≤ 2.5 x ULN.
12. Adequate cardiac function with left ventricular ejection fraction ≥ 50% by echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan.

    * QTc interval ≤ 460 ms using Fredericia's QT correction formula (at baseline from ECGs). NOTE: Participants with a right or left bundle branch block are allowed to have a QTc > 460ms.
    * Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class I or II and stage A or B
13. For dose expansion cohort: the participant must be willing to undergo biopsy procedure at screening and on treatment.

Exclusion Criteria

1. Participants who are pregnant or lactating.
2. Participants with sarcoma components of their endometrial cancer, except carcinosarcoma.
3. Radiation, chemotherapy, or immunotherapy or any other anticancer therapy ≤2 weeks prior to cycle 1 day 1.
4. Participation in an interventional anti-cancer study (clinical trial) within 3 weeks prior to cycle 1 day 1
5. Major surgery within four weeks before cycle 1 day 1.
6. A history of congestive heart failure (CHF) of NYHA Class ≥3, or history of myocardial infarction (MI) within 3 months.
7. Participants with a history of severe obstructive pulmonary disease, pulmonary hypertension, and/or pulmonary fibrosis in the opinion of treating MD
8. History of medically significant rhabdomyolysis in the opinion of treating MD.
9. For participants with prior MEK inhibitors, any history of or ongoing Grade 4 toxicity deemed related to MEK inhibitor
10. Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; participants with controlled infection in the opinion of treating MD or on prophylactic antibiotics are permitted in the study.
11. Hepatitis B, or C infection as indicated by detectable viral load. Known to be HIV seropositive with detectable viral load. Participants with an undetectable viral load are eligible for the trial.
12. Any underlying condition that would significantly interfere with the absorption of an oral medication or inability to take oral medications in the opinion of treating MD
13. Participants with psychiatric illness/social situations that would limit compliance with study requirements.
14. Participants with symptomatic brain lesions
15. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation). Subjects with known deep vein thrombosis/pulmonary embolism that are under appropriate anti-coagulation treatment are eligible
16. History of clinically significant hemoptysis within 1 month prior to study enrollment for any tumor type.
17. Current, non-healing wound, ulcer or bone fractures
18. Known hypersensitivity to defactinib, avutometinib, everolimus, and/or other rapamycin derivatives.
19. Current warfarin use. Participants who are being treated with warfarin within 7-14 days prior to enrollment for deep vein thrombosis/pulmonary embolism may be eligible if their warfarin therapy can be converted to low molecular weight heparin or direct oral anticoagulants (DOACs). Participants who can be transitioned should have INR checked after 5 days on low molecular weight heparin or a direct oral anticoagulant (DOAC).

    Participants are eligible if the INR is ≤ 1.5 prior to the first study dose.
20. Current use of medications (with or without prescriptions), supplements, herbal remedies, or foods (Grapefruit and grapefruit juice, Seville oranges and star fruit) with potential for drug-drug interactions with avutometinib and/or defactinib within 5 half-lives (if known), or if not known then 14 days prior to the first dose of study intervention, including:

    * Strong CYP3A4 inhibitors or inducers
    * Strong CYP2C9 inhibitors or inducers
    * Strong P-glycoprotein (P-gp) inhibitors or inducers
    * Strong breast cancer resistance protein (BCRP) inhibitors or inducers
21. Specific concurrent ocular disorders:

    * History of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes
    * History of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mmHg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
    * Active or chronic, visually significant corneal disorders, other active ocular conditions requiring ongoing therapy, or clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy. Examples of visually significant corneal disorders include corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions. Visually significant corneal disorders do NOT include dry eyes, blepharitis, and uncomplicated corneal erosions.
22. Severe skin disorder in the opinion of treating MD that has required systemic therapy within one year of the first dose of study intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2026-06-03 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs). | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org